CLINICAL TRIAL: NCT03523962
Title: PREPARE: A Pragmatic Randomized Trial Evaluating Pre-operative Alcohol Skin Solutions in FRactured Extremites
Brief Title: Pre-operative Alcohol Skin Solutions in Fractured Extremities
Acronym: PREPARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: McMaster University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Gerard Slobogean, Assistant Professor, Department of Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00080639
Record Dates: First submitted 2018-04-30; First posted 2018-05-14 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Surgical Site Infection; Unplanned Fracture-Related Reoperation; Open Appendicular Fracture; Closed Lower Extremity Fracture; Pelvic Fracture
Keywords: Surgical Site Infection; Open Fracture; Lower Extremity Fracture; Pelvis; Fracture; DuraPrep; ChloraPrep; Peri-operative Preparation Solutions
MeSH Terms: conditions — Surgical Wound Infection; Hip Fractures; Fractures, Open | interventions — DuraPrep

STUDY DESIGN:
Intervention Model Description: Treatment allocation will be determined using a cluster-randomized crossover trial design. The open and closed fracture populations will be treated with the same allocated solution at all times during the trial. The order of treatment allocation for each orthopaedic practice will be randomly assigned using a computer-generated randomization table. Each site will start with the initially allocated study solution and eventually crossover to the other solution for their second recruitment period. This process of alternating treatments will repeat approximately every 2 months as dictated by the initial randomization.
Who Masked: Outcomes Assessor
Masking Description: The orthopaedic team (including the study coordinators) cannot be blinded to the treatment allocation as the antiseptic solutions are visually distinguishable and these individuals need to lead the implementation of the cluster-crossover protocol at their clinical site. The Adjudication Committee Members and data analysts will be blinded to the study treatment. All interpretation of study results will initially be done in a blinded manner by developing two interpretations of the results. One interpretation will assume treatment A is iodine povacrylex, the other interpretation will assume it is CHG. Once the data interpretations for each assumption are finalized, the data will be unblinded and the correct interpretation will be accepted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- First pre-op antiseptic skin solution (Experimental): The PREPARE trial will compare the most common alcohol-based pre-operative antiseptic skin solutions used during extremity fracture surgery. Participant recruitment will begin with the clinical sites using their assigned pre-operative antiseptic skin solution for all eligible fracture surgeries for a two-month period.
  Interventions: Drug: DuraPrep; Drug: ChloraPrep
- Crossover - Second pre-op antiseptic skin solution (Experimental): Once the first intervention phase is completed, each site will crossover to the opposite study solution. Each site will need to develop local procedures to ensure a successful crossover. They will use the second solution for all eligible fracture surgeries for a two-month period, and will then crossover back to the solution in the first intervention phase.
  Interventions: Drug: DuraPrep; Drug: ChloraPrep

INTERVENTIONS:
Drug: DuraPrep — The iodine-based treatment intervention is an antiseptic solution comprised of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol. 3M™ DuraPrep™ [3M Health Care, St Paul, MN], will be the commercial product used.
Drug: ChloraPrep — The CHG intervention is an antiseptic solution comprised of 2% CHG in 70% isopropyl alcohol. ChloraPrep® [CareFusion Inc., Leawood, KS, USA] will be the product used.

SUMMARY:
The prevention of infection is an important goal influencing peri-operative care of extremity fracture patients. Standard practice in the operative management of extremity fractures includes sterile technique and pre-operative skin preparation with an antiseptic solution. The available solutions kill bacteria and decrease the quantity of native skin flora, thereby decreasing surgical site infection (SSI). While there is extensive guidance on specific procedures for prophylactic antibiotic use and standards for sterile technique, the evidence regarding the choice of antiseptic skin preparation solution is very limited for extremity fracture surgery.

DETAILED DESCRIPTION:
More than one million Americans suffer an extremity fracture (broken bone in the arm, leg, or pelvis) that requires surgery each year. Approximately 5% (or 50,000) of surgical fracture patients develop a surgical site infection (SSI), which is twice the rate among most surgical patients and nearly five times the rate among patients undergoing elective orthopaedic surgeries (e.g. joint replacement). Patients who develop a SSI after their fracture fixation surgery experience a long and difficult treatment pathway. Researchers have identified that when a fracture patient experiences a SSI, they typically undergo at least two additional surgeries to control the infection, spend a median of 14 additional days in the hospital, and have significantly lower health related quality of life (HRQL). Similarly, results from the recently completed Fluid Lavage of Open Wounds (FLOW) trial confirmed that patients who had a SSI, or another complication, that required an additional surgery reported significantly lower physical and mental HRQL in the 12 months following their fracture compared to patients who did not experience a SSI. In the most severe cases, when a SSI cannot be controlled, a limb amputation becomes necessary.

Open fractures, closed lower extremity fractures, and pelvic fractures represent some of the most severe musculoskeletal injuries. Due to their high-energy mechanisms, these fractures are often accompanied by soft-tissue injuries that contribute to unacceptably poor outcomes. The FLOW trial of 2,447 open fracture patients reported a 13.2% incidence of open fracture-related reoperations; Closed fractures of the lower extremity are also at high risk of complications, particularly when compared to closed upper extremity fractures. For example, the rate of SSI in closed tibial plateau and plafond fractures range from 5.6 - 11.9%, although some cohort studies have reported infection rates as high as 25.0%. This is contrast with SSI rates of <5% for common upper extremity fractures like humeral shaft, forearm, or distal radius fractures. This is further illustrated in a series of 214 deep orthopaedic fracture infections, in which 58% occurred in the tibia and ankle, and only 10% occurred anywhere in the upper extremity. Finally, pelvic fractures are associated with some of the most challenging SSIs to treat among closed fractures because of their propensity to gram negative organisms and limitations in reconstruction options post-infection. Ultimately, infectious complications in these fracture populations lead to prolonged morbidity, loss of function, and potential limb loss.

ELIGIBILITY:
The open fracture inclusion criteria are:

1. Patients 18 years of age or older.
2. Open fracture of the appendicular skeleton.
3. Received or will receive definitive fracture treatment with a surgical implant(s) (i.e., internal fixation, external fixation, joint prosthesis, etc.).
4. Open fracture wound management that includes formal surgical debridement within 72 hours of their injury.
5. Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
6. Informed consent obtained.
7. Patient enrolled within 3 weeks of their fracture.

The open fracture exclusion criteria are:

1. Fracture of the hand (distal to radial carpal joint).
2. Patients who did not or will not receive the allocated pre-operative surgical preparation solution due to a medical contraindication.
3. Received previous surgical debridement or management of their fracture at a nonparticipating hospital or clinic (as applicable).
4. Open fracture managed outside of the participating orthopaedic service (e.g., foot fracture managed by podiatrist).
5. Chronic or acute infection at or near the fracture site at the time of initial fracture surgery.
6. Burns at the fracture site.
7. Incarceration.
8. Expected injury survival of less than 90 days.
9. Terminal illness with expected survival less than 90 days.
10. Currently enrolled in a study that does not permit co-enrollment.
11. Unable to obtain informed consent due to language barriers.
12. Likely problems, in the judgment of study personnel, with maintaining follow-up with the patient.
13. Prior or current enrollment in a PREP-IT trial.
14. Enrolled in the PREPARE closed cohort.
15. Excluded due to sampling strategy.

The closed fracture inclusion criteria are:

1. Patients 18 years of age or older.
2. Closed fracture of the lower extremity or pelvis.
3. Received or will receive definitive fracture treatment with a surgical implant(s) (i.e., internal fixation, external fixation, joint prosthesis, etc.).
4. Fracture management requires a surgical incision (i.e., for fracture reduction or implant insertion).
5. Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
6. Informed consent obtained.
7. Patient enrolled within 6 weeks of their fracture.

The closed fracture exclusion criteria are:

1. Patients who did not or will not receive the allocated pre-operative surgical preparation solution due to a medical contraindication.
2. Received previous surgical management of their fracture at a non-participating hospital or clinic.
3. Fracture managed outside of the participating orthopaedic service (e.g., foot fracture managed by podiatrist).
4. Chronic or acute infection at or near the fracture site at the time of initial fracture surgery.
5. Burns at the fracture site.
6. Incarceration.
7. Expected injury survival of less than 90 days.
8. Terminal illness with expected survival less than 90 days.
9. Currently enrolled in a study that does not permit co-enrollment.
10. Unable to obtain informed consent due to language barriers.
11. Likely, problems, in the judgment of study personnel, with maintaining follow-up with the patient.
12. Prior or current enrollment in a PREP-IT trial.
13. Enrolled in the PREPARE open cohort.
14. Excluded due to sampling strategy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8485 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Slobogean, MD, Principal Investigator — University of Maryland, Baltimore; Sheila Sprague, PhD, Principal Investigator — McMaster University; Mohit Bhandari, MD, Principal Investigator — McMaster University
Locations (27):
- United States (24):
  - University of California, Irvine, Irvine, California
  - Cedars Sinai, Los Angeles, California
  - Regional Medical Center of San Jose, San Jose, California
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Louisiana State University, Baton Rouge, Louisiana
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - University of Maryland Capital Region Health, Cheverly, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Bryan Health, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Hanover, New Hampshire
  - Carolinas Medical Center, Atrium Health Musculoskeletal Institute, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest Baptist University Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Case Western / MetroHealth Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - San Antonio Military Medical Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Health System Foundation / Inova Fairfax Hospital, Falls Church, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Canada (3):
  - Royal Columbia Hospital, New Westminster, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - McMaster University, Center for Evidence-Based Orthopaedics, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] PREP-IT Investigators; Sprague S, Slobogean G, Wells JL, O'Hara NN, Thabane L, Mullins CD, Harris AD, Wood A, Viskontas D, Apostle KL, O'Toole RV, Joshi M, Johal H, Al-Asiri J, Hymes RA, Gaski GE, Pilson HT, Carroll EA, Babcock S, Halvorson JJ, Romeo NM, Matson CA, Higgins TF, Marchand LS, Bergin PF, Morellato J, Van Demark RE 3rd, Potter GD, Gitajn IL, Chang G, Phelps KD, Kempton LB, Karunakar M, Jaeblon T, Demyanovich HK, Domes CM, Kuhn GR, Reilly RM, Gage MJ, Weaver MJ, von Keudell AG, Heng M, McTague MF, Alnasser A, Mehta S, Donegan DJ, Natoli RM, Szatkowski J, Scott AN, Shannon SF, Jeray KJ, Tanner SL, Marmor MT, Matityahu A, Fowler JT, Pierrie SN, Beltran MJ, Thomson CG, Lin CA, Moon CN, Scolaro JA, Amirhekmat A, Leonard J, Pogorzelski D, Bzovsky S, Heels-Ansdell D, Szasz OP, Gallant JL, Della Rocca GJ, Zura RD, Hebden JN, Patterson JT, Lee C, O'Hara LM, Marvel D, Palmer JE, Friedrich J, D'Alleyrand JG, Rivera JC, Mossuto F, Schrank GM, Guyatt G, Devereaux PJ, Bhandari M; The PREP-IT Investigators. Skin Antisepsis before Surgical Fixation of Extremity Fractures. N Engl J Med. 2024 Feb 1;390(5):409-420. doi: 10.1056/NEJMoa2307679. PMID 38294973
- [Derived] Boissonneault A, O Hara N, Pogorzelski D, Marchand L, Higgins T, Gitajn L, Gage MJ, Natoli RM, Sharma I, Pierrie S, O'Toole RV, Sprague S, Slobogean G; PREP-IT Investigators*. The impact of heterotopic ossification prophylaxis after surgical fixation of acetabular fractures: national treatment patterns and related outcomes. Injury. 2023 Mar 6:S0020-1383(23)00197-3. doi: 10.1016/j.injury.2023.03.001. Online ahead of print. PMID 37002119
- [Derived] Sprague S, Scott T, Dodds S, Pogorzelski D, McKay P, Harris AD, Wood A, Thabane L, Bhandari M, Mehta S, Gaski G, Boulton C, Marcano-Fernandez F, Guerra-Farfan E, Hebden J, O'Hara LM, Slobogean GP; PREP-IT Investigators. Cluster identification, selection, and description in cluster randomized crossover trials: the PREP-IT trials. Trials. 2020 Aug 12;21(1):712. doi: 10.1186/s13063-020-04611-9. PMID 32787892
- [Derived] Program of Randomized Trials to Evaluate Pre-operative Antiseptic Skin Solutions in Orthopaedic Trauma (PREP-IT) Investigators; Slobogean GP, Sprague S, Wells J, Bhandari M, Rojas A, Garibaldi A, Wood A, Howe A, Harris AD, Petrisor BA, Mullins DC, Pogorzelski D, Marvel D, Heels-Ansdell D, Mossuto F, Grissom F, Del Fabbro G, Guyatt GH, Della Rocca GJ, Demyanovich HK, Gitajn IL, Palmer J, D'Alleyrand JC, Friedrich J, Rivera J, Hebden J, Rudnicki J, Fowler J, Jeray KJ, Thabane L, Marchand L, O'Hara LM, Joshi MG, Talbot M, Camara M, Szasz OP, O'Hara NN, McKay P, Devereaux PJ, O'Toole RV, Zura R, Morshed S, Dodds S, Li S, Tanner SL, Scott T, Nguyen U. Effectiveness of Iodophor vs Chlorhexidine Solutions for Surgical Site Infections and Unplanned Reoperations for Patients Who Underwent Fracture Repair: The PREP-IT Master Protocol. JAMA Netw Open. 2020 Apr 1;3(4):e202215. doi: 10.1001/jamanetworkopen.2020.2215. PMID 32259266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between August 21, 2018, and March 18, 2023 at 25 hospitals in the United States and Canada. Of these hospitals, 20 recruited patients with either open or closed fractures; 3 hospitals recruited patients with closed fractures only, and 2 recruited those with open fractures only.
Pre-assignment Details: To ensure wide generalizability to routine practice, the protocol allowed prewashing of the operative extremity with alcohol or other antiseptics before performing the final skin antisepsis with the study solution. In addition to ensuring trial feasibility and protocol adherence, this decision pragmatically allowed the intact skin to receive mechanical scrubbing or partial alcohol antisepsis at the treating surgeon's discretion.
Units Other Than Participants: Clinical Sites
Groups:
- Closed Fractures - Iodine Povacrylex First, Then Chlorhexidine Gluconate: The closed-fracture population consisted of adults (≥18 years old) who were undergoing surgical fixation of a closed lower-limb or pelvic fracture. We excluded patients who had a concurrent open fracture, had a medical contraindication to receive either trial intervention, or had a chronic or acute infection at or near the fracture site at the time of the index surgery.
  The iodine-based treatment intervention is an antiseptic solution comprised of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol. 3M™ DuraPrep™ [3M Health Care, St Paul, MN], was the commercial product used.
  The CHG intervention is an antiseptic solution comprised of 2% CHG in 70% isopropyl alcohol. ChloraPrep® [CareFusion Inc., Leawood, KS, USA] was the product used.
- Closed Fractures - Chlorhexidine Gluconate First, Then Iodine Povacrylex: The closed-fracture population consisted of adults (≥18 years old) who were undergoing surgical fixation of a closed lower-limb or pelvic fracture. We excluded patients who had a concurrent open fracture, had a medical contraindication to receive either trial intervention, or had a chronic or acute infection at or near the fracture site at the time of the index surgery.
  The CHG intervention is an antiseptic solution comprised of 2% CHG in 70% isopropyl alcohol. ChloraPrep® [CareFusion Inc., Leawood, KS, USA] was the product used.
  The iodine-based treatment intervention is an antiseptic solution comprised of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol. 3M™ DuraPrep™ [3M Health Care, St Paul, MN], was the commercial product used.
- Open Fractures - Iodine Povacrylex First, Then Chlorhexidine Gluconate: The open-fracture population consisted of adults (≥18 years old) who had an open upper-limb or lower-limb fracture warranting surgical fixation. In addition, the patient's open fracture must have received surgical débridement within 72 hours after injury. We excluded patients with open fractures of the hand and those who had received previous surgical debridement at a nonparticipating hospital.
  The iodine-based treatment intervention is an antiseptic solution comprised of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol. 3M™ DuraPrep™ [3M Health Care, St Paul, MN], was the commercial product used.
  The CHG intervention is an antiseptic solution comprised of 2% CHG in 70% isopropyl alcohol. ChloraPrep® [CareFusion Inc., Leawood, KS, USA] will be the product used.
- Open Fractures - Chlorhexidine Gluconate First, Then Iodine Povacrylex: The open-fracture population consisted of adults (≥18 years old) who had an open upper-limb or lower-limb fracture warranting surgical fixation. In addition, the patient's open fracture must have received surgical débridement within 72 hours after injury. We excluded patients with open fractures of the hand and those who had received previous surgical debridement at a nonparticipating hospital.
  The CHG intervention is an antiseptic solution comprised of 2% CHG in 70% isopropyl alcohol. ChloraPrep® [CareFusion Inc., Leawood, KS, USA] was the product used.
  The iodine-based treatment intervention is an antiseptic solution comprised of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol. 3M™ DuraPrep™ [3M Health Care, St Paul, MN], will be the commercial product used.
Period: Closed Fractures
Arm/Group | Closed Fractures - Iodine Povacrylex First, Then Chlorhexidine Gluconate | Closed Fractures - Chlorhexidine Gluconate First, Then Iodine Povacrylex | Open Fractures - Iodine Povacrylex First, Then Chlorhexidine Gluconate | Open Fractures - Chlorhexidine Gluconate First, Then Iodine Povacrylex
Started | 2748; 12 Clinical Sites | 4037; 11 Clinical Sites | 0; 0 Clinical Sites | 0; 0 Clinical Sites
Iodine Povacrylex | 1405; 12 Clinical Sites | 1955; 11 Clinical Sites | 0; 0 Clinical Sites | 0; 0 Clinical Sites
Chlorhexidine Gluconate | 1343; 12 Clinical Sites | 2082; 11 Clinical Sites | 0; 0 Clinical Sites | 0; 0 Clinical Sites
Completed | 2580; 12 Clinical Sites | 3897; 11 Clinical Sites | 0; 0 Clinical Sites | 0; 0 Clinical Sites
Not Completed | 168; 0 Clinical Sites | 140; 0 Clinical Sites | 0; 0 Clinical Sites | 0; 0 Clinical Sites
Not completed — Death | 86 | 71 | 0 | 0
Not completed — Lost to Follow-up | 62 | 36 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 29 | 0 | 0
Not completed — Incarceration | 1 | 4 | 0 | 0
Period: Open Fractures
Arm/Group | Closed Fractures - Iodine Povacrylex First, Then Chlorhexidine Gluconate | Closed Fractures - Chlorhexidine Gluconate First, Then Iodine Povacrylex | Open Fractures - Iodine Povacrylex First, Then Chlorhexidine Gluconate | Open Fractures - Chlorhexidine Gluconate First, Then Iodine Povacrylex
Started | 0; 0 Clinical Sites | 0; 0 Clinical Sites | 987; 11 Clinical Sites | 713; 11 Clinical Sites
Iodine Povacrylex | 0; 0 Clinical Sites | 0; 0 Clinical Sites | 503; 11 Clinical Sites | 351; 11 Clinical Sites
Chlorhexidine Gluconate | 0; 0 Clinical Sites | 0; 0 Clinical Sites | 484; 11 Clinical Sites | 362; 11 Clinical Sites
Completed | 0; 0 Clinical Sites | 0; 0 Clinical Sites | 954; 11 Clinical Sites | 697; 11 Clinical Sites
Not Completed | 0; 0 Clinical Sites | 0; 0 Clinical Sites | 33; 0 Clinical Sites | 16; 0 Clinical Sites
Not completed — Death | 0 | 0 | 11 | 6
Not completed — Lost to Follow-up | 0 | 0 | 15 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 2
Not completed — Incarceration | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Closed-Fracture Population Iodine Group: The closed-fracture population consisted of adults (≥18 years old) who were undergoing surgical fixation of a closed lower-limb or pelvic fracture. We excluded patients who had a concurrent open fracture, had a medical contraindication to receive either trial intervention, or had a chronic or acute infection at or near the fracture site at the time of the index surgery.
  The iodine-based treatment intervention is an antiseptic solution comprised of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol. 3M™ DuraPrep™ [3M Health Care, St Paul, MN], will be the commercial product used.
- Closed-Fracture Population Chlorhexidine Group: The closed-fracture population consisted of adults (≥18 years old) who were undergoing surgical fixation of a closed lower-limb or pelvic fracture. We excluded patients who had a concurrent open fracture, had a medical contraindication to receive either trial intervention, or had a chronic or acute infection at or near the fracture site at the time of the index surgery.
  The CHG intervention is an antiseptic solution comprised of 2% CHG in 70% isopropyl alcohol. ChloraPrep® [CareFusion Inc., Leawood, KS, USA] will be the product used.
- Open-Fracture Population Iodine Group: The open-fracture population consisted of adults (≥18 years old) who had an open upper-limb or lower-limb fracture warranting surgical fixation. In addition, the patient's open fracture must have received surgical débridement within 72 hours after injury. We excluded patients with open fractures of the hand and those who had received previous surgical debridement at a nonparticipating hospital.
  The iodine-based treatment intervention is an antiseptic solution comprised of iodine povacrylex (0.7% free iodine) in 74% isopropyl alcohol. 3M™ DuraPrep™ [3M Health Care, St Paul, MN], will be the commercial product used.
- Open-Fracture Population Chlorhexidine Group: The open-fracture population consisted of adults (≥18 years old) who had an open upper-limb or lower-limb fracture warranting surgical fixation. In addition, the patient's open fracture must have received surgical débridement within 72 hours after injury. We excluded patients with open fractures of the hand and those who had received previous surgical debridement at a nonparticipating hospital.
  The CHG intervention is an antiseptic solution comprised of 2% CHG in 70% isopropyl alcohol. ChloraPrep® [CareFusion Inc., Leawood, KS, USA] will be the product used.
- Total: Total of all reporting groups
Arm/Group | Closed-Fracture Population Iodine Group | Closed-Fracture Population Chlorhexidine Group | Open-Fracture Population Iodine Group | Open-Fracture Population Chlorhexidine Group | Total
Number analyzed (Participants) | 3360 | 3425 | 854 | 846 | 8485
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (20.2) | 53.6 (20.4) | 45.0 (18.3) | 44.2 (18.1) | 47.0 (19.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 1730 | 1739 | 312 | 309 | 4090
  Sex: Male | 1629 | 1686 | 542 | 537 | 4394
  Sex: Missing Data | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 170 | 181 | 65 | 47 | 463
  Not Hispanic or Latino | 3190 | 3244 | 789 | 799 | 8022
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 2652 | 2706 | 584 | 589 | 6531
  Race: Black | 501 | 480 | 227 | 214 | 1422
  Race: Asian | 140 | 147 | 22 | 17 | 326
  Race: Indigenous | 27 | 33 | 9 | 12 | 81
  Race: Central or South American | 4 | 7 | 2 | 1 | 14
  Race: Multiracial | 3 | 4 | 2 | 4 | 13
  Race: Native Hawaiian or Pacific Islander | 3 | 5 | 1 | 1 | 10
  Race: Missing Data | 30 | 43 | 7 | 8 | 88
BMI [Count of Participants; unit: Participants]
  Underweight (<18.5 kg/m^2) | 99 | 80 | 12 | 13 | 204
  Healthy weight (18.5 - 24.9 kg/m^2) | 1068 | 1106 | 252 | 250 | 2676
  Overweight (25.0-29.9 kg/m^2) | 1082 | 1024 | 279 | 294 | 2679
  Obesity (>30.0 kg/m^2) | 1111 | 1215 | 311 | 289 | 2926
Diabetes of any type [Count of Participants; unit: Participants] | 470 | 445 | 80 | 64 | 1059
Current smoker [Count of Participants; unit: Participants] | 753 | 722 | 289 | 282 | 2046
Injury Severity Score (ISS) [Mean (Standard Deviation); unit: units on a scale] — An established medical score to assess trauma severity. To calculate, take the highest severity code (1=Minor, 2=Moderate, 3=Serious, 4=Severe, 5=Critical, 6=Unsurvivable) in each of the three most severely injured ISS body regions (Head, Face, Chest, Abdomen, Extremity, External), square each code and add the three squared numbers (ISS = A2 + B2 + C2 where A, B, C are the severity codes of the three most injured ISS body regions). ISS ranges from 1 to 75. If any of the three scores is a 6, the score is automatically set at 75.
  units on a scale | 9.0 (6.2) | 8.9 (6.2) | 13.4 (8.5) | 12.9 (8.0) | 11.1 (7.2)
American Society of Anesthesiologist (ASA) Physical Score [Count of Participants; unit: Participants] — The American Society of Anesthesiologist (ASA) score is a subjective assessment of a patient's overall health that is based on five classes (I to V).
  I. Patient is a completely healthy fit patient. II. Patient has mild systemic disease. III. Patient has severe systemic disease that is not incapacitating. IV. Patient has incapacitating disease that is a constant threat to life. V. A moribund patient who is not expected to live 24 hour with or without surgery.
  Participants
    Class I or II | 1760 | 1752 | 440 | 463 | 4415
    Class III or higher | 1600 | 1673 | 414 | 383 | 4070
Number of included fractures per participant [Count of Participants; unit: Participants]
  One | 3169 | 3240 | 782 | 771 | 7962
  Two | 166 | 162 | 62 | 68 | 458
  Three | 25 | 23 | 10 | 7 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Superficial Incisional Surgical Site Infection (SSI)
Description: Guided by the Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network reporting criteria (2017):
  Date of event for infection may occur from the date of fracture to 30 days after the definitive fracture management surgery; AND involves only skin and subcutaneous tissue of the incision; AND patient has at least one of the following:
  1. purulent drainage from the superficial incision.
  2. organisms identified from an aseptically obtained specimen from the superficial incision or subcutaneous tissue by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment
  3. superficial incision that is deliberately opened by a surgeon, and culture or non-culture-based testing is not performed. AND patient has at least one of the following signs or symptoms: pain or tenderness; localized swelling; erythema; or heat.
  4. diagnosis of a superficial incisional SSI by the surgeon.
Time Frame: Within 30 days of the patient's last planned fracture management surgery
Population: Outcome data for surgical-site infection were missing for 4.5% of the patients in the closed-fracture population and for 2.8% of those in the open-fracture population.
Measure: Count of Participants; unit: Participants
Arm/Group | Closed-Fracture Population Iodine Group | Closed-Fracture Population Chlorhexidine Group | Open-Fracture Population Iodine Group | Open-Fracture Population Chlorhexidine Group
Number analyzed (Participants) | 3205 | 3272 | 825 | 826
Participants | 20 | 27 | 6 | 9

2. Primary Outcome: Number of Participants With a Deep Incisional Infection
Description: Guided by CDC's National Healthcare Safety Network Surgical Site Infection reporting criteria (2017):
  Deep Incisional Infection:
  Occurs within 90 days post definitive fracture management; & involves fascial/muscle layers; & has at least one of the following:
  1. deep incision purulent drainage
  2. a deep incision that dehisces, or is opened by a surgeon, and organism is identified by microbiologic testing; or microbiologic testing is not performed & has at least one of the following: fever (> 38 °C); localized pain or tenderness
  3. other evidence of deep incision infection on anatomical exam or imaging test
Time Frame: Within 90 days of the patient's last planned fracture management surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Closed-Fracture Population Iodine Group | Closed-Fracture Population Chlorhexidine Group | Open-Fracture Population Iodine Group | Open-Fracture Population Chlorhexidine Group
Number analyzed (Participants) | 3205 | 3272 | 825 | 826
Participants | 29 | 54 | 21 | 20

3. Secondary Outcome: Number of Participants With an Unplanned Fracture-Related Reoperation
Description: Common examples include any unplanned fracture-related surgery that is associated with an infection at the operative site or contiguous to it, a wound-healing problem, or a fracture delayed union or non-union.
Time Frame: Within 12 months of the patient's last planned operation
Population: Primary and secondary outcomes were evaluated using a complete case analysis. For that reason, the overall number of participants analyzed differs from the numbers provided under the Participant Flow module.
Measure: Count of Participants; unit: Participants
Arm/Group | Closed-Fracture Population Iodine Group | Closed-Fracture Population Chlorhexidine Group | Open-Fracture Population Iodine Group | Open-Fracture Population Chlorhexidine Group
Number analyzed (Participants) | 2982 | 3047 | 784 | 785
Participants | 164 | 179 | 126 | 114

ADVERSE EVENTS:
Time Frame: 1 year post injury
Description: This study did not collect data regarding "Other (Not Including Serious) Adverse Events".
Arm/Group | Closed-Fracture Population Iodine Group | Closed-Fracture Population Chlorhexidine Group | Open-Fracture Population Iodine Group | Open-Fracture Population Chlorhexidine Group
All-Cause Mortality (participants affected / at risk) | 145/3360 | 140/3425 | 13/854 | 13/846
Serious Adverse Events (participants affected / at risk) | 1177/3360 | 1212/3425 | 430/854 | 368/846
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed-Fracture Population Iodine Group (N=3360) | Closed-Fracture Population Chlorhexidine Group (N=3425) | Open-Fracture Population Iodine Group (N=854) | Open-Fracture Population Chlorhexidine Group (N=846)
Study Fracture Related Complication (Musculoskeletal and connective tissue disorders) | 347 (347) | 360 (360) | 198 (198) | 187 (187)
Non-Study Fracture Related Complication (Musculoskeletal and connective tissue disorders) | 33 (33) | 36 (36) | 40 (40) | 26 (26)
Neurological (Nervous system disorders) | 33 (33) | 34 (34) | 3 (3) | 10 (10)
Renal (Renal and urinary disorders) | 81 (81) | 82 (82) | 22 (22) | 16 (16)
Cardiac (Cardiac disorders) | 88 (88) | 90 (90) | 16 (16) | 6 (6)
Vascular (Vascular disorders) | 43 (43) | 41 (41) | 15 (15) | 12 (12)
Gastro-Intestinal (Gastrointestinal disorders) | 58 (58) | 59 (59) | 21 (21) | 7 (7)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 93 (93) | 90 (90) | 29 (29) | 21 (21)
Other (General disorders) | 401 (401) | 420 (420) | 86 (86) | 83 (83)

LIMITATIONS AND CAVEATS:
1. The patients and their surgeons were aware of the trial-group assignments.
2. The trial was limited to patients undergoing surgery for a fracture, so the generalizability of these findings to other surgical populations is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT03523962/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03523962/SAP_001.pdf